CLINICAL TRIAL: NCT03931460
Title: Feasibility of Medical Abortion by Telemedicine in Mexico
Status: Completed | Type: Observational
Sponsor: Gynuity Health Projects (Other)
Responsible Party: Sponsor
Other Study IDs: 1045
Record Dates: First submitted 2019-04-25; First posted 2019-04-30 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Pregnancy
MeSH Terms: interventions — Abortion, Induced

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Medical Abortion — Medical Abortion
  Other Names: Medication abortion, abortion with pills

SUMMARY:
This study is designed to obtain preliminary data on the safety, acceptability, and feasibility of direct-to-consumer telemedicine abortion in Mexico.

DETAILED DESCRIPTION:
This is a case-series prospective study to develop, implement, and evaluate a telemedicine medical abortion service in private sector health facilities in Mexico. The service will be designed to incorporate the standard steps in an in-person medical abortion procedure, thus ensuring that the quality of care provided to each woman is equal to that which she would receive if she presented in person to an abortion facility.

Individuals determined as likely to be eligible will have a "TelEvaluation" by videoconference, telephone, messaging, or a combination of these, with a study provider who will give standard pre-abortion counseling and explain study procedures and the process of obtaining informed consent for the study. The informed consent form will be either signed electronically using secure software, or by printing the form, signing, scanning, and returning it to the study site; oral consent recorded by telephone will be also an option. Demographic and medical information will be recorded during the TelEvaluation. If required by the site, the provider will assist in identifying facilities to obtain any tests and have the results sent to the study site.

A person will be eligible for the study if they have no contraindications to medical abortion medications, if an intrauterine pregnancy is determined, and if the provider judge that the participant could receive and take the mifepristone at ≤70 days of gestation. If the individual is eligible and wishes to continue with the abortion, the site will send a package containing one tablet of mifepristone 200 mg, 8 tablets of misoprostol 200 mcg, and 8 tablets of ibuprofen 800 mg once payment for the service is received. Each site will determine the total cost of the service, and the package will be shipped by tracked mail or other reliable means of delivery. Distance to the clinic will be measured using a map application and the address provided by the participant for package receipt. Antibiotics, antiemetics, and contraceptives will be prescribed at the discretion of the site. The package will also include written instructions detailing medication administration, expected symptoms and side effects, the follow up plan, and emergency procedures. The regimen to be used is mifepristone 200 mg followed by misoprostol 800 mcg within 48 h administered buccally or sublingually. The participant will be instructed to take the remaining four misoprostol tablets if no bleeding occurred within 24 hours of taking the misoprostol dose.

A follow-up contact with the study provider will be scheduled for 7 to 14 days after the package is mailed to assess abortion outcome, adverse events, and other relevant information via phone interview or messaging. Study providers will use any combination of methods to determine abortion completeness including ultrasound, serum HCG, urine pregnancy test, and patient's history. If further care is indicated, the provider will refer the participant to a facility. Once it is found that the abortion is complete staff will administer a satisfaction questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Woman is pregnant and desires a medical abortion by remote consult (TeleAborto)
* Woman has access to internet or equipment for a remote consult
* Woman can provide address to which abortifacient medications will be mailed
* Woman reports no contraindications to medical abortion
* The study site does not suspect an ectopic pregnancy or nonviable pregnancy
* The gestational age allows sufficient time for the woman to take the mifepristone on or before 70 days of gestation
* A feasible plan is made that the woman agrees to confirm complete abortion and to seek care to manage incomplete abortion complications
* The woman understands and is likely to comply with study instructions and has granted informed consent to participate in the study.

Exclusion Criteria:

* Medically ineligible for procedure.

Ages: 10 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Women seeking abortion
Sampling Method: Non-Probability Sample
Enrollment: 1114 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability | 1 year
  Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Beverly B Winikoff, MD, MPH, Principal Investigator — Gynuity Health Projects
Locations (5):
- Mexico (5):
  - Telefem, Mexico City, Mexico City
  - Atención Integral en Ginecología,Medieg A.C., Mexico City
  - Centro de Atención Integral a la Pareja, A.C. (CIPA), Mexico City
  - Gineclinic, Mexico City
  - MUSOR, Oaxaca City